CLINICAL TRIAL: NCT03539705
Title: Food Allergy Registry at a Single Site
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Food Allergy Research & Education (Other)
Responsible Party: Principal Investigator, R. Sharon Chinthrajah, MD, Associate Professor, Stanford University
Other Study IDs: 36273; 1UM1AI130839-01 (NIH); 1U01AI182039-01 (NIH)
Record Dates: First submitted 2018-05-16; First posted 2018-05-29 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Allergy and Asthma
MeSH Terms: conditions — Hypersensitivity; Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: There is no intervention — There is no intervention

SUMMARY:
This is a registry of participants who are interested in being screened for clinical trials at a single site.

DETAILED DESCRIPTION:
This registry will be maintained on a secure database and will include demographics information such as name, gender, age, date of birth, ethnicity, race, and contact information, disease, medical information, other information (via questionnaires), and date of consent. It will be overseen by our data manager at our site and will not be shared with others outside of our site-specific trained individuals.

ELIGIBILITY:
Inclusion Criteria:

* Any interested party from 0-100 yrs of age to enter their information in registry

Exclusion Criteria:

* Any individual who does not consent

Ages: 0 Years to 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Any interested party from 0-100 yrs of age to enter their information in registry
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2018-01-05 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Registry to provide a list of interested individuals in clinical trials at a single site | 4 years
  The clinical trials could be either allergy or asthma studies

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Chinthrajah, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No